CLINICAL TRIAL: NCT00173719
Title: Influence of Assistive Device Use on Dynamic Balance and the Associated Attentional Demands During Standing and Walking in Patients With Stroke
Brief Title: Influence of Assistive Device Use While Performing Dual Task in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 9100002423
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-01

CONDITIONS: Stroke
Keywords: Hemiplegia; Assisstive device; Walking; Dynamic equilibrium; Reaction time; Attention; Dual task
MeSH Terms: conditions — Stroke; Hemiplegia

INTERVENTIONS:
Device: Standard cane

SUMMARY:
The primary purposes of the this three-year research proposal are to investigate the influence of assistive device use on dynamic balance and the associated attentional demands during standing and walking in patients with stroke

DETAILED DESCRIPTION:
Research has shown the effectiveness of using ambulatory assistive devices to increase standing stability of patients with stroke in clinical practice (Maeda et al., 2001). However, literature has also suggested that manipulation of ambulatory assistive devices in dynamic motor tasks, such as walking, inevitably requires additional attention, even in healthy adults (Wright & Kemp, 1992). Given that the majority of patients with stroke suffer from balance control difficulty, which subsequently increases their attentional demands associated with maintaining balance (Brown et al., 2002), it remains an important question as to whether the use of ambulatory assistive devices would take away some attentional resources that would otherwise be used for maintaining balance.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults

* between 50 and 75 years old
* having no neuromuscular or musculoskeletal disorders that would jeopardize their balance control abilities
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital

Stroke patients

* between 50 and 75 years old
* hemiplegic or hemiparetic as a result of a single cerebral vascular accident
* medically stable with no ongoing complications
* independently walking without using any assistive device for at least 10 meters, and have the exercise endurance for at least 30 minutes
* having no serious hemianopsia, hemi-inattention or any obvious cognitive problems as evaluated with the Mini-Mental State examination
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital

Exclusion Criteria:

* unable to follow the order of the experimenters, and having serious comprehension and expression impairment

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-09; Primary Completion 2004-01 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To investigate the voice reaction time and response accuracy while simultaneously performing the dual task with or without using assistive devices for healthy adults and stroke patients | 2003-2004

SECONDARY OUTCOMES:
To investigate the related gait parameters(ex. walking speed, stride length, gait cycle time, and foot pressure etc.)while simultaneously performing the dual task with or without using assistive devices for healthy adults and stroke patients

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Taiwan